CLINICAL TRIAL: NCT00772265
Title: A Randomized Single Center Double Blind 2 Period Crossover Glucose Clamp Study to Test for Bioequivalence Between 2 Recombinant Human Isophane Insulins Wockhardt's Human Isophane Insulin Injection100IU/ml With Novolin N in Healthy Subjects
Brief Title: Comparative Glucose Clamp Study of Wockhardt's Human Isophane Insulin With Novolin N,in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wockhardt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: WosulinN/PK-PD/HV/FDA/10/v3
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-12

CONDITIONS: Diabetes
Keywords: Bioequivalence; pharmacokinetic; Pharmacodynamic; Isophane insulin
MeSH Terms: conditions — Diabetes Mellitus | interventions — Isophane Insulin, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wosulin N (Experimental): Wosulin N, Isophane insulin for injection (Recombinant Human Insulin)(100 IU/mL), cartridges 3.0 mL
  Interventions: Biological: Wosulin N
- Novolin N (Active Comparator): Novolin N, Isophane insulin for injection (Recominant Human Insulin)(100IU/ml),cartridges 3.0ml.
  Interventions: Biological: Novolin N

INTERVENTIONS:
Biological: Wosulin N — Total Dose per subject will be 0.4IU/Kg given Subcutaneously.
  Arms: Wosulin N
Biological: Novolin N — Total dose per subject will be 0.4 IU/Kg given Subcutaneously.
  Arms: Novolin N

SUMMARY:
The aim of this trial is to demonstrate bioequivalence of Wosulin N to Novolin® N with regard to its total and to its maximum serum insulin concentrations.

DETAILED DESCRIPTION:
The purpose of this study is is to test for bioequivalence based on AUC0-24h and Cmax between Wosulin N and Novolin® N.The study also compares the pharmacokinetic and pharmacodynamic profiles as well as assessing safety and local tolerability of the two insulin preparations in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subject.
* Age more than 18 and less than 45 years.
* Considered generally healthy upon completion of medical history, physical examination and biochemical investigations as judged by the Investigator.
* Body Mass Index (BMI) between 18.0 and 27.0 kg/m2, inclusive.
* Non-smoker, defined as no nicotine consumption for at least one year.
* Signed and dated informed consent obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the subject.)

Exclusion Criteria:

* Previous participation in this trial or other clinical trials within the last 30 days.
* Pregnant, breast-feeding or intention of becoming pregnant or not using adequate contraceptive measures (defined as intrauterine device (IUD) that has been in place for at least 3 months, double barrier contraception, sterilization or abstinence, or oral contraceptive pill, which should have been taken without difficulty for at least 3 months, or an approved hormonal implant).
* Clinically significant abnormal haematology or biochemistry screening tests, as judged by the Investigator. In particular, subjects with elevated liver enzymes (AST or ALT > 2 times the upper limit of normal) or impaired renal function (elevated serum creatinine values above the upper limit of normal) will not be allowed to enter the trial.
* Any serious systemic infectious disease during the four weeks prior to the first dose of test drug, as judged by the Investigator.
* History of any illness that, in the opinion of the Investigator, might confound the results of the trial or pose risk in administering the trial drug to the subject. In particular, subjects with significant cardiovascular disease, anemia (haemoglobin below the lower limit of normal) or hemoglobinopathy will not be allowed to enter the trial.
* History of alcohol or drug abuse in the past five years and/or any positive test for drugs of abuse at screening.
* Any positive reaction of drugs of abuse.
* Hepatitis B or C or HIV positive.
* Use of prescription drugs within 3 weeks preceding the first dosing of insulin, except for oral contraceptives/hormonal implants.
* Use of any insulin product for therapeutic purposes in the past.
* Use of non-prescription drugs, except routine vitamins, within 3 weeks prior to the first dose of the test drug. Occasional use of acetaminophen is permitted.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or co-operation.
* Blood donation of more than 500 ml within the last 12 weeks.
* History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction.
* Known or suspected allergy to trial product or related products.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2010-09; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Mean AUC0-24h and Cmax | Visit 2 and 3

SECONDARY OUTCOMES:
PK endpts: AUC0-4h, AUC0-6h, AUC0-12h, AUC6-12h, AUC6-24h,tmax,and elimination rate constant. PD endpoints: AUCGIR0-4h, AUCGIR0-6h, AUCGIR0-12h,AUCGIR0-24h, AUCGIR6-12h, AUCGIR6-24h, GIRmax and tGIRmax Safety : AEs,haematology,biochem,phy exam. | Visit 2,3 and 4

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Guthrie, Study Chair — Profil Institute for Clinical Research, Inc.
Locations (1):
- Profil Institute for clinical Research, Chula Vista, California, United States